CLINICAL TRIAL: NCT03391635
Title: Efficacy of Electroacupuncture Compared With Transcutaneous Electric Nerve Stimulation for Functional Constipation:a Randomized Controlled Trial
Brief Title: Efficacy of Electroacupuncture Compared With Transcutaneous Electric Nerve Stimulation for Functional Constipation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Yuxiao Zeng, Postgraduate student of China Academy of Chinese Medical Sciences, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GAMHospital20171222
Record Dates: First submitted 2017-12-22; First posted 2018-01-05 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Functional Constipation
Keywords: acupuncture; functional constipation; transcutaneous electric nerve stimulation; randomized controlled trial
MeSH Terms: interventions — Electroacupuncture; Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electroacupuncture (Experimental): The treatment consists of 3 times a week for 8 weeks.Huatuo Brand needles (0.30×50mm or 0.30×70mm) and the SDZ-V EA apparatus (Suzhou Medical Appliance) will be used for ST25, SP14 and ST37.After acupuncture，the needle handle will be connected with the electrode in the electroacupuncture instrument.
  The parameters of the electric acupuncture apparatus：Dilatational wave，the frequency is 2/10Hz，the electric current intensity is 0.1mA-1.0mA.
  Interventions: Device: Electroacupuncture
- TranscutaneousElectricNerveStimulation (Active Comparator): The treatment consists of 3 times a week for 8 weeks.Huatuo Brand electrode patch (50mm×50mm) and the SDZ-V EA apparatus (Suzhou Medical Appliance) will be used for ST25, SP14 and ST37.
  The parameters of the electric acupuncture apparatus：Dilatational wave，the frequency is 2/10Hz，the electric current intensity is 2mA-5mA.
  Interventions: Device: TranscutaneousElectricNerveStimulation

INTERVENTIONS:
Device: Electroacupuncture — Participants will receive electroacupuncture at bilateral ST25, SP14 and ST37 for 30 minutes each time，3 times a week for 8 weeks.
  Other Names: EA
  Arms: Electroacupuncture
Device: TranscutaneousElectricNerveStimulation — Participants will receive transcutaneous electric nerve stimulation at bilateral ST25, SP14 and ST37 for 30 minutes each time，3 times a week for 8 weeks.
  Other Names: TENS
  Arms: TranscutaneousElectricNerveStimulation

SUMMARY:
The objective of this trial is to compare the efficacy of electroacupuncture versus transcutaneous electric nerve stimulation for functional constipation

DETAILED DESCRIPTION:
Both electroacupuncture(EA) therapy and transcutaneous electric nerve stimulation(TENS) are safe and effective for functional constipation, but no head to head comparing trial was conducted.

Methods：102 participants with functional constipation will be recruited and randomly allocated into the EA group and the TENS group.Participants in both groups will receive EA or TENS treatment at Tianshu(ST 25), Fujie(SP 14) and Shangju xu(ST 37) 3 times a week for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Conforming to the criteria for the diagnosis of functional constipation in Rome III standard;
2. Aged of 18 to 75 years;
3. No medication for constipation has been used for at least 2 weeks before treatment. Except for emergency treatment, it has not received acupuncture treatment for constipation in the past 3 months, and has not participated in other ongoing clinical research.

Exclusion Criteria:

1. Constipation caused by irritable bowel syndrome and organically or medicated; secondary to endocrine, metabolic, neurogenic, or surgical constipation;
2. Subjects with serious heart, liver, kidney damage or cognitive impairment, aphasia, mental disorders, or the inability to cooperate with the examination and treatment.
3. Pregnant or lactation patients;
4. Subjects with abdominal aortic aneurysm, abnormal enlargement of liver and spleen and so on.
5. Subjects with coagulation dysfunction or anticoagulants such as warfarin and heparin have been used all the time.
6. Subjects installed with the cardiac pacemaker.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
The proportion of participants with an average increasing of one or more complete spontaneous bowel movements from baseline at week 8. | Baseline，week 8
  The proportion of participants with an average increasing of one or more complete spontaneous bowel movements from baseline at week 8.

SECONDARY OUTCOMES:
The proportion of participants with an average increasing of one or more complete spontaneous bowel movements | Baseline，week 4，week 20 and week 32
  The proportion of participants with an average increasing of one or more complete spontaneous bowel movements from baseline at weeks 4 , 20 and 32.
Change number in CSBMS | Baseline，week 4，week 8, week 20 and week 32
  The change in the number of CSBMs at weeks 4 , 8 , 20 and 32.
Change number in SBMS | Baseline，week 4，week 8, week 20 and week 32
  The change in the number of SBMs at weeks 4 , 8 , 20 and 32.
The proportion of participants with type3 or type 4 stool character | Baseline，week 4，week 8, week 20 and week 32
  According to the BRISTOL stool form scale, the proportion of participants with type3 or type 4 at weeks 4 , 8 , 20 and 32
Change number of average score in defecation difficulty | Baseline，week 4，week 8, week 20 and week 32
  The change in average score of difficulty in defecation at weeks 4 , 8 , 20 and 32
Change number of PAC-QOL score | Baseline，week 8
  The change in total score on the patients assessment of constipation quality of life questionnaire(PAC-QOL) total score at the end of week 8, compared with baseline.
The proportion and average amount of using cathartics | weeks -1 , 4 , 8 , 20 and 32.
  The proportion and average amount of using cathartics at weeks -1 , 4 , 8 , 20 and 32.

CONTACTS AND LOCATIONS:
Overall Officials: Yuxiao Zeng, Principal Investigator — Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Locations (1):
- Guang'anmen Hospital of China Academy of Chinese Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mugie SM, Benninga MA, Di Lorenzo C. Epidemiology of constipation in children and adults: a systematic review. Best Pract Res Clin Gastroenterol. 2011 Feb;25(1):3-18. doi: 10.1016/j.bpg.2010.12.010. PMID 21382575
- [Result] Tran LC, Di Palma JA. Lack of lasting effectiveness of PEG 3350 laxative treatment of constipation. J Clin Gastroenterol. 2005 Aug;39(7):600-2. doi: 10.1097/01.mcg.0000170769.67320.47. PMID 16000928
- [Result] Gordon M, Naidoo K, Akobeng AK, Thomas AG. Osmotic and stimulant laxatives for the management of childhood constipation. Cochrane Database Syst Rev. 2012 Jul 11;(7):CD009118. doi: 10.1002/14651858.CD009118.pub2. PMID 22786523
- [Result] Pare P, Bridges R, Champion MC, Ganguli SC, Gray JR, Irvine EJ, Plourde V, Poitras P, Turnbull GK, Moayyedi P, Flook N, Collins SM. Recommendations on chronic constipation (including constipation associated with irritable bowel syndrome) treatment. Can J Gastroenterol. 2007 Apr;21 Suppl B(Suppl B):3B-22B. PMID 17464377
- [Result] Ford AC, Suares NC. Effect of laxatives and pharmacological therapies in chronic idiopathic constipation: systematic review and meta-analysis. Gut. 2011 Feb;60(2):209-18. doi: 10.1136/gut.2010.227132. PMID 21205879
- [Result] Wong SW, Lubowski DZ. Slow-transit constipation: evaluation and treatment. ANZ J Surg. 2007 May;77(5):320-8. doi: 10.1111/j.1445-2197.2007.04051.x. PMID 17497967
- [Result] Pfeifer J. Surgical options to treat constipation: A brief overview. Rozhl Chir. 2015 Sep;94(9):349-61. PMID 26537099
- [Result] Remes Troche JM, Gomez Escudero O, Icaza Chavez ME, Noble Lugo A, Lopez Colombo A, Bielsa MV, Charua Guindic L; Asociacion Mexicana de Gastroenterologia. [Guidelines for diagnosis and treatment of constipation in Mexico. C) Medical and surgical treatment]. Rev Gastroenterol Mex. 2011 Apr-Jun;76(2):141-54. Spanish. PMID 21724490
- [Result] Du WF, Yu L, Yan XK, Wang FC. [Met-analysis on randomized controlled clinical trials of acupuncture and moxibustion on constipation]. Zhongguo Zhen Jiu. 2012 Jan;32(1):92-6. Chinese. PMID 22295840
- [Result] Liu Z, Yan S, Wu J, He L, Li N, Dong G, Fang J, Fu W, Fu L, Sun J, Wang L, Wang S, Yang J, Zhang H, Zhang J, Zhao J, Zhou W, Zhou Z, Ai Y, Zhou K, Liu J, Xu H, Cai Y, Liu B. Acupuncture for Chronic Severe Functional Constipation: A Randomized Trial. Ann Intern Med. 2016 Dec 6;165(11):761-769. doi: 10.7326/M15-3118. Epub 2016 Sep 13. PMID 27618593
- [Result] Drossman DA. The functional gastrointestinal disorders and the Rome III process. Gastroenterology. 2006 Apr;130(5):1377-90. doi: 10.1053/j.gastro.2006.03.008. No abstract available. PMID 16678553
- [Result] Lewis SJ, Heaton KW. Stool form scale as a useful guide to intestinal transit time. Scand J Gastroenterol. 1997 Sep;32(9):920-4. doi: 10.3109/00365529709011203. PMID 9299672
- [Result] Marquis P, De La Loge C, Dubois D, McDermott A, Chassany O. Development and validation of the Patient Assessment of Constipation Quality of Life questionnaire. Scand J Gastroenterol. 2005 May;40(5):540-51. doi: 10.1080/00365520510012208. PMID 16036506
- [Result] Yang X, Liu Y, Liu B, He L, Liu Z, Yan Y, Liu J, Liu B. Factors related to acupuncture response in patients with chronic severe functional constipation: Secondary analysis of a randomized controlled trial. PLoS One. 2017 Nov 22;12(11):e0187723. doi: 10.1371/journal.pone.0187723. eCollection 2017. PMID 29166673
- [Result] Ismail KA, Chase J, Gibb S, Clarke M, Catto-Smith AG, Robertson VJ, Hutson JM, Southwell BR. Daily transabdominal electrical stimulation at home increased defecation in children with slow-transit constipation: a pilot study. J Pediatr Surg. 2009 Dec;44(12):2388-92. doi: 10.1016/j.jpedsurg.2009.07.063. PMID 20006033
- [Result] Clarke MC, Chase JW, Gibb S, Hutson JM, Southwell BR. Improvement of quality of life in children with slow transit constipation after treatment with transcutaneous electrical stimulation. J Pediatr Surg. 2009 Jun;44(6):1268-72; discussion 1272. doi: 10.1016/j.jpedsurg.2009.02.031. PMID 19524752